CLINICAL TRIAL: NCT01244451
Title: A Single-Arm Multi-Center Trial of Bendamustine Given With Ofatumumab (BendOfa) in Patients With Refractory or Relapsed Chronic Lymphocytic Leukemia (CLL). EudraCT Number 2009-017663-42. GIMEMA CLL0809 Protocol
Brief Title: GIMEMA CLL0809 Study (BendOfa)
Acronym: BendOfa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL0809
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Patients With CLL Relapsing After an Initial Response (CR, PR ≥ 6 Months) Following no More Than Two Prior Treatment Lines; or; Patients With CLL Refractory (SD, PD or CR/PR < 6 Months) Following no More Than Two Prior Treatment Lines
Keywords: CLL; relapsed; refractory; Bendamustine; Ofatumumab
MeSH Terms: conditions — Recurrence | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendofa (Experimental): Bendamustine + Ofatumumab
  Interventions: Drug: Ofatumumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab will be administered at the dose of 300 mg IV D1 and 1000 mg IV D8 1st course; 1000 mg IV D1, 2nd -6th courses.
Drug: Bendamustine — Bendamustine will be infused at the doses of 70 mg/m2 IV on days D1 and D2 of each course.

SUMMARY:
In the last ten years there have been significant developments in CLL treatment. The advent of fludarabine, rituximab and the association of chemo-immunotherapy have substantially increased overall response rate, CR rate, time to progression and may also have an impact on overall survival.

Even though, CLL remains incurable and all patients eventually relapse and progressively become resistant to treatment. The development of an effective therapy that is not cross-resistant with the ones currently available as front-line treatment, is one of the clinical unmet needs within CLL.

BendOfa is a non comparative phase II trial designed to determine the therapeutic benefit of bendamustine given together to ofatumumab in relapsed or resistant patients with CLL.

Bendamustine is approved by FDA for CLL treatment, it is an hybrid drug with alkylating agents and purine analogue properties that may lack of cross resistance with fludarabine. It was utilized in CLL as a single agent and its association with rituximab is currently under clinical investigation.

Ofatumumab is a new fully human anti-CD20 monoclonal antibody with high in vitro efficacy on CD20 low-expressing CLL cells. An early report showed that ofatumumab in single therapy is effective in highly pre-treated refractory CLL patients.

Both drugs were generally well tolerated without unexpected untoward toxicity. On the basis of these data, bendamustine and ofatumumab could be a new effective and well tolerated combination for patients with relapsed and refractory CLL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL relapsing after an initial response (CR, PR ≥ 6 months) following no more than two prior treatment lines; or
* Patients with CLL refractory (SD, PD or CR/PR < 6 months) following no more than two prior treatment lines
* Patients requiring treatment according to 2008 revised IWCLL guidelines
* No more than 2 prior treatment lines
* Age older or equal to 18 years
* No active malignancies during the previous 5 years, with the exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of any origin
* No prior treatment with conventional chemotherapy within the prior 4 weeks and with monoclonal antibodies within the prior 16 weeks
* ECOG performance status of ≤2 at study entry
* Laboratory test results within these ranges:

Serum creatinine ≤ 2 x UNL Creatinine clearance ≥ 50 ml/min (Cockcroft and Gault formula) Total bilirubin ≤ 2 x UNL (with exception of patients with Gilbert's syndrome) AST (SGOT) and ALT (SGPT) ≤ 2 x UNL non attributable to CLL AST (SGOT) and ALT (SGPT) ≤ 10 x UNL attributable to CLL

* Female subjects of childbearing potential(FCBP) must:

Understands the potential teratogenic risk to the unborn child and the need for effective contraception;

Be capable of complying with effective contraceptive measures.

Be informed and understand the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy.

Understand the need to commence the study treatment as soon as study drug is dispensed following a negative pregnancy test.

Understand the need and accepts to undergo pregnancy testing based on the frequency outlined in this protocol.

Females of childbearing potential (FCBP) enrolled in this protocol must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation.

The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:

Highly effective methods:

* Intrauterine device (IUD)
* Hormonal (birth control pills, injections, implants)
* Tubal ligation
* Partner's vasectomy

Additional effective methods:

* Male condom
* Diaphragm
* Cervical Cap
* Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia.
* Pregnancy testing.

FCBP must have two negative pregnancy tests prior to starting study drug.

FCBP must agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.

Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.

- Male patients must:

Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a female of childbearing potential.

Must practice complete abstinence or agree to use a prophylactic during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 6 months following study drug discontinuation, even if he has undergone a successful vasectomy.

If pregnancy or a positive pregnancy test does occur in the partner of a male study patient during study participation, the investigator must be notified immediately.

- Female and male patients

should be instructed never to give this medicinal product to another person and to return any unused capsules to the study doctor at the end of treatment.

Should not donate blood during therapy and for at least 28 days following discontinuation of study drug.

Male patients should not donate semen or sperm while participating in the study, during dose interruptions and for at least 6 months following study drug discontinuation

* Signed written informed consent according to IGH/EU/GCP and Italian laws.

Exclusion Criteria:

* Concurrent use of other anti-cancer agents
* Use of any other experimental drug or therapy within 28 days of baseline
* Positive direct antiglobulin test (DAT) with clinical and laboratory signs of hemolysis and/or autoimmune thrombocytopenia
* Known transformation of CLL
* Known CNS involvement of CLL
* Known positivity for HIV or active HCV and HBV hepatitis.
* Active bacterial, viral or fungal infection requiring systemic anti-viral, antibiotic or anti-fungal therapy.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones or stable chronic liver disease per investigator assessment)
* Pregnant or Lactating Females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she was to participate in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Cortelezzi, Pr., Principal Investigator — Direzione Scientifica - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena
Locations (32):
- Italy (32):
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - Azienda Sanitaria di Bolzano - Ospedale Centrale - Ematologia e Centro TMO, Bolzano
  - Azienda ASL di Cagliari, Cagliari
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Clinica Ematologica - Università degli Studi, Genova
  - ASL Le1 P.O. Vito Fazzi - U.O. di Ematologia, Lecce
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Messina Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - Sez. di medicina Interna Oncologia ed Ematologia, Modena
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Dipartimento Emato-Oncologia A.O. "Bianchi-Melacrino-Morelli", Reggio Calabria
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Università degli studi di Roma La Cattolica, Roma
  - Ospedale S.Eugenio, Rome
  - Ospedale Casa Sollievo della sofferenza, San Giovanni Rotondo
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - SS.C. di Oncoematologia - Dipartimento di Medicina Clinica e Sperimentale - Azienda Ospedaliera - S. Maria Di Terni, Terni
  - Div. di Ematologia "Molinette" Osp. Maggiore S. G. Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Policlinico G.B. Rossi, Verona

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it/en/index.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bendofa
Started | 49
Completed | 36
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Bendofa
Number analyzed (Participants) | 49
Age, Continuous [Mean (Full Range); unit: Years] | 65.85 [46.12 to 81.18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Contributing to the Overall Response Rate
Description: Patients response to treatment will be assessed by clinical examination, peripheral blood, bone marrow aspirate and biopsy and radiographic evaluation according to the revised IWCLL 2008 criteria.
Time Frame: After 8 months from therapy start (6 months of treatment plus 2 months from the last course to response evaluation)
Measure: Number; unit: participants
Arm/Group | Bendofa
Number analyzed (Participants) | 44
participants | 34

2. Secondary Outcome: Toxicity According to CTCAE Version 4.0
Description: Number of patients experiencing 3 or >3 AEs (both hematological and not hematological)
Time Frame: At 44 months from treatment start.
Population: Number of patients experiencing 3 or >3 Adverse Events (AEs) (both hematological and not hematological)
Measure: Number; unit: participants
Groups:
- Study Group: Number of patients experiencing 3 or >3 AEs (both hematological and not hematological)
Arm/Group | Study Group
Number analyzed (Participants) | 49
participants | 47

3. Secondary Outcome: Progression Free Survival
Description: Patients still alive and known to be progression-free will be censored at the moment of last follow-up. Patients disease progression will be assessed by clinical examination, peripheral blood, bone marrow aspirate and biopsy and radiographic evaluation according to the revised IWCLL 2008 criteria.
Time Frame: Up to 32 months: from the date of first BendOfa treatment dose - induction phase - until the date of the first documentation of progressive disease or until death (whatever the cause), whichever occurs first.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendofa
Number analyzed (Participants) | 49
Participants | 49

4. Secondary Outcome: Overall Survival
Description: Patients still alive will be censored at the moment of last follow-up.
Time Frame: At 44 months from treatment start.
Measure: Number; unit: participants
Arm/Group | Bendofa
Number analyzed (Participants) | 47
participants | 38

ADVERSE EVENTS:
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 47/49
Other Adverse Events (participants affected / at risk) | 19/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=49)
Anemia (Blood and lymphatic system disorders) | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 22
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=49)
Vomiting (Gastrointestinal disorders) | 2
Allergic dermatitis (Blood and lymphatic system disorders) | 1
Allergic reaction (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cough (General disorders) | 1
Dyspnoea (General disorders) | 1
Fatigue (General disorders) | 2
Gastrointestinal hemorrhage (General disorders) | 1
Hypotension (General disorders) | 2
Nausea (General disorders) | 2
Other toxicity (General disorders) | 3
Rash (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs of participating centres may disclose their centre's results only after the main study publication has been released, so that a single centre experience can be compared to the study overall results and give a more appropriate view of the study.